CLINICAL TRIAL: NCT06406309
Title: Settling Down for Sleep: The Impact of Sensory and Arousal Systems on Sleep in ADHD
Brief Title: Settling Down for Sleep in ADHD: The Impact of Sensory and Arousal Systems on Sleep in ADHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: The Klingenstein Third Generation Foundation (Other)
Responsible Party: Principal Investigator, Amy Hartman, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24030096
Record Dates: First submitted 2024-05-01; First posted 2024-05-09 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Attention Deficit Hyperactivity Disorder; Sleep Disturbance
Keywords: Sleep disturbances; Emotion Dysregulation; Sensory Processing; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Parasomnias

STUDY DESIGN:
Intervention Model Description: Micro-longitudinal (3 weeks total, daily measurement) observational baseline (1 week) and 2 week intervention study trialing a bedtime manipulation intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Settle down to sleep (Experimental): All participants will engage in a 1 week home-based baseline measurement, 1 lab visit for training and measurement, and 2 week intervention trial.
  Interventions: Behavioral: Power Down manipulation

INTERVENTIONS:
Behavioral: Power Down manipulation — The Power Down is a bedtime manipulation protocol targeting elevated arousal level at bedtime due to a hypothesized effect of sensory over-responsivity (a common experience for children with ADHD). The Power Down incorporates sensory-based tools (gentle tactile pressure and auditory cues) to support nervous system regulation prior to attempting sleep onset. Caregivers will lead a nightly gentle massage with guided relaxation script just prior to the child trying to fall asleep during the 2-week intervention phase. The child will also wear a watch-like activity monitor (ActiGraph GT9x) for the 2 week period throughout the day and night to measure changes in sleep and activity patterns. Caregivers will complete daily diary questions in the morning and evening reporting their child's emotions and sleep timing.

SUMMARY:
The goal of this study is test the hypothesis that sleep problems for children with ADHD are linked to sensory over-responsivity, a type of sensory processing difference that causes a person to interpret daily sensory input as stressful. This study examines the impact of sensory over-responsivity on bedtime arousal levels in 30 children with ADHD (ages 6-13). We will also test a bedtime intervention targeting sensory over-responsivity at bedtime and examine how it impacts bedtime arousal levels and sleep difficulties.

DETAILED DESCRIPTION:
Following the consent process, baseline data collection will be completed electronically with questionnaires sent digitally to participants (parent and child) using a secure, web-based application (REDCap). Participants will then complete a virtual clinical baseline interview and training on the wear of the EmbracePlus ("watch") and the daily virtual sleep diary. Upon completion of this, the study team will then send the watch and its accessories to the participant via the mail.

Time point 1 home-based data collection (1 week): Once the caregiver and child receive the watch and study materials, home-based data collection will start. During this 1-week period, the child will wear the watch 24-hours/day for one week and the caregiver(s) will complete daily sleep diary entries (morning and evening). At the end of this data collection period, the study materials will be brought into the lab session.

Lab-based session (1-2 hours): Participants and caregivers will complete a training session on the environmental changes and a novel bedtime manipulation intervention called the "Power Down".

Time point 2 home-based data collection (2 weeks): Participants will apply any sleep environment changes identified during the lab session, complete the 'power down" each night, child will wear the watch 24hrs/day, and caregivers will complete daily sleep diaries (morning and evening). At the end of this timepoint, all study materials will be mailed back to the study team and a virtual exit interview will be completed. Final sleep and intervention acceptability questionnaires will be completed virtually.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 6-13 years
* A reported clinical diagnosis of ADHD or suspected ADHD and 6+ items endorsed as "quite a bit" or "very much" a single domain on SNAP-IV (ADHD symptomology questionnaire)
* Parents endorse >20 minutes to settle down and fall asleep
* Caregiver willing to participate in all bedtimes during intervention.
* Willing to come into the lab in Pittsburgh

Exclusion Criteria:

* Concurrent organic sleep disorder (sleep apnea, narcolepsy), psychiatric (major depression, bipolar, OCD, psychosis, schizophrenia)
* Current behavioral treatment for sleep disorder
* Unstable ADHD medication use (dose or timing)
* Children who have trauma or other histories for whom physical touch is triggering (per caregiver report) will be excluded.
* If a child spends bedtime at a different caregiver's home for >50% of the nights and that caregiver is not willing to participate in this study, the child will be excluded from this study.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
General Sensory over-responsivity | Baseline
  Caregiver-reported Sensory Profile-2 questionnaire: Sensitivity sub scale score (score range of 0 - 95, with higher numbers indicating more frequent endorsement)
General bedtime arousal | Baseline
  Pre-Sleep Arousal Scale total score (range of 16-80): caregiver- and child-reported arousal experiences prior to bedtime. Likert scale (1-5, with 1 indicating that the person does not experience the symptom at all and 5 indicating that a person experiences the symptom extremely).
General Emotion dysregulation | Baseline
  Emotion Dysregulation Inventory Short Form: Reactivity and Dysphoria total scores: Caregiver-reported questionnaire scored on a Likert scale from 1 ("Not at all") to 5 (Very Severe"). Reactivity sub scale is a total of 8 questions (range of 8-40) and dysphoria sub scale is a total of 5 questions (range of 5-25).
Daily bedtime arousal level | Daily for 2 weeks
  The Empatica Embrace Plus is a watch-like device that captures movement and electrodermal activity during wear. The child will wear the Empatica all day and night for 2 weeks. The bedtime period will be isolated and measures of movement (maximum magnitude of activity using accelerometery) and electrodermal activity (maximum skin conductance levels) will be extracted to assess bedtime arousal level nightly.
Daily bedtime emotion dysregulation | Daily for 2 weeks
  Emotion Dysregulation Inventory Short Form Reactivity and Dysphoria sub scales: Caregiver-reported questionnaire scored on a Likert scale from 1 ("Not at all") to 5 (Very Severe"). Reactivity sub scale is a total of 8 questions (range of 8-40) and dysphoria sub scale is a total of 5 questions (range of 5-25).
Change in sleep disturbances | Baseline and after 2 week intervention
  Change in PROMIS Sleep Disturbances Scale: Caregiver reported outcome with 15 questions on a Likert scale of 1 ("Never") to 5 ("Always"). Scoring ranges from 15 - 75. Baseline and post intervention total scores will be examined to measure change in sleep disturbances across time.
Intervention Feasibility | After 2 week intervention
  Feasibility of Intervention Measure (FIM): Caregiver-reported questionnaire with 4 questions on a Likert scale of 1 ("Completely disagree") to 5 ("Completely agree"). Scoring ranges from 4-20.
Intervention Acceptability | After 2 week intervention
  Acceptability of Intervention Measure (AIM): Caregiver-reported questionnaire with 4 questions on a Likert scale of 1 ("Completely disagree") to 5 ("Completely agree"). Scoring ranges from 4-20.
Intervention Appropriateness | After 2 week intervention
  Intervention Appropriateness Measure (IAM): Caregiver-reported questionnaire with 4 questions on a Likert scale of 1 ("Completely disagree") to 5 ("Completely agree"). Scoring ranges from 4-20.

SECONDARY OUTCOMES:
Circadian preference | Baseline
  Morningness and Eveningness Questionnaire: Child-reported questionnaire with 10 multiple choice questions scored on a scale of 1 to 4 or 5 with a higher score indicating a stronger morning preference and a lower score indicating minimal morning preference (range of score is 10 - 42)
Change in sleep difficulties | Daily across 2 weeks
  Using the actigraphy data and data from daily diaries, we will calculate sleep onset latency each night of baseline (1 week) and across the 1 week of intervention trial
Change in sleep related impairment | Baseline and after 2 week intervention
  Change in total score of the PROMIS Sleep Related Impairment Scale: Caregiver reported outcome with 4 questions on a Likert scale of 1 ("Never") to 5 ("Always"). Scoring ranges from 4-20. Total score will be collected at baseline and post intervention and change scores will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Amy G Hartman, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The full study protocol and informed consent forms will be shared with interested researchers upon request. Only aggregate and de-identified data collected throughout the clinical trial will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available to share after publication of findings or 2 years after the end of the study, whichever comes first.
Access Criteria: Data will be shared with researchers within and outside of the University of Pittsburgh through email requests to the lead principal investigator. The University of Pittsburgh may require a data use agreement be developed and signed by both institutions.